CLINICAL TRIAL: NCT05477056
Title: Quality Improvement Survey I.0: A Retrospective Data Analysis of Clinician Survey Responses Following the Utilization of the PrecivityADTM Blood Test for the Detection of Alzheimer's Disease Pathology (QUIP I)
Brief Title: Quality Improvement PrecivityAD Clinician Survey (QUIP I)
Acronym: QUIP I
Status: Completed | Type: Observational
Sponsor: C2N Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: C2N001
Record Dates: First submitted 2022-07-23; First posted 2022-07-28 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Dementia; Cognitive Decline
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PrecivityAD blood test — Clinician Survey post receipt of PrecivityAD blood test result
  Other Names: AD

SUMMARY:
There is an important unmet need for timely, non-invasive, and low-burden evaluation of patients presenting with mild cognitive impairment (MCI) and early dementia. MCI impacts 12-18% of people in the United States over age 60 and is often an initial clinical sign of Alzheimer's disease (AD) (Alzheimer's Association, 2022). The PrecivityAD test is an analytically and clinically validated blood test that aids healthcare providers in the diagnosis of AD in patients with MCI and early-stage dementia. C2N has created a quality improvement (QI) survey to gather insight from clinicians as to the clinical effectiveness of the commercially available PrecivityAD™ test, which identifies whether a patient with signs and symptoms of cognitive decline is likely to have amyloid plaques in the brain, a pathological hallmark of Alzheimer's disease.

DETAILED DESCRIPTION:
By gathering feedback from healthcare providers on patient selection, intended use, and anticipated outcomes and continued or revised care plans as a result of the test report, C2N can better understand the impact of the test results on diagnosis and patient management.

ELIGIBILITY:
Inclusion Criteria:

1. Memory specialist actively practicing in the United States.
2. Practice includes individuals with mild cognitive impairment age > 60 years
3. Average patient volume > 50 visits per week (all patients seen across practice)

Exclusion Criteria:

1. Other clinicians with a specialty outside of the field of Memory Specialists
2. Principal Investigator reserves the right to not include a clinician in the survey

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Memory Specialists actively practicing in the United States were asked to complete the QI 1.0 survey with expertise in caring for patients with mild cognitive impairment and knowledge of Alzheimer's Disease in terms of expertise and volume of patients served. This may include nurse practitioners or physician assistants who work in the field of Memory Disorders.
Sampling Method: Non-Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
evaluate patient selection for the blood test through analysis of clinician survey responses. | 2021 - 2023
  retrospective analysis of clinician survey data collected during a single timepoint
evaluate score interpretation for the Amyloid Probability Score (APS) through analysis of clinician survey responses. | 2021 - 2023
  retrospective analysis of clinician survey data collected during a single timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Tim West, Ph.D, Principal Investigator — C2N
Locations (1):
- C2N Diagnostics, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monane M, Johnson KG, Snider BJ, Turner RS, Drake JD, Maraganore DM, Bicksel JL, Jacobs DH, Ortega JL, Henderson J, Jiang Y, Huang S, Coppinger J, Fogelman I, West T, Braunstein JB. A blood biomarker test for brain amyloid impacts the clinical evaluation of cognitive impairment. Ann Clin Transl Neurol. 2023 Oct;10(10):1738-1748. doi: 10.1002/acn3.51863. Epub 2023 Aug 7. PMID 37550958